CLINICAL TRIAL: NCT00475501
Title: 5-Alpha Reductase and Anabolic Effects of Testosterone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Endo Pharmaceuticals (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDA-014-05F; VA Merit Award (Other Grant/Funding Number: VHA AR6884R)
Record Dates: First submitted 2007-04-16; First posted 2007-05-21 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Male Hypogonadism; Muscle Atrophy; Sarcopenia; Benign Prostate Hypertrophy
Keywords: anabolic effects; finasteride; male hypogonadism; sarcopenia; testosterone
MeSH Terms: conditions — Eunuchism; Muscular Atrophy; Sarcopenia; Prostatic Hyperplasia | interventions — testosterone enanthate; Finasteride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): testosterone enanthate
  Interventions: Drug: Testosterone Enanthate
- Arm 2 (Experimental): finasteride
  Interventions: Drug: Finasteride
- Arm 3 (Experimental): testosterone enanthate + finasteride
  Interventions: Drug: Testosterone Enanthate; Drug: Finasteride
- Arm 4 (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Testosterone Enanthate — 125 mg, i.m. injection, once/week, for 52 weeks
  Other Names: Delatestryl
  Arms: Arm 1; Arm 3
Drug: Finasteride — 5 mg, oral, once/day, for 52 weeks
  Other Names: Proscar
  Arms: Arm 2; Arm 3
Other: Placebo — Placebo
  Arms: Arm 4

SUMMARY:
The purpose of this study is to determine whether a higher-than-replacement dose of testosterone and finasteride can be combined to safely increase muscle strength in older men who have a low blood concentration of testosterone.

DETAILED DESCRIPTION:
Approximately 40% of older male veterans have a low serum testosterone concentration. The latter is associated with diminished muscle strength and bone mineral density, depressed mood, low pain tolerance, frailty, and increased mortality. Replacement doses of testosterone have been administered to hypogonadal men for the purpose of reversing deficits in muscle and bone. Although testosterone is clearly important for maintaining muscle and bone in men, there are problems associated with T replacement. First, testosterone causes a number of undesired effects, including fluid retention, gynecomastia, worsening of sleep apnea, polycythemia, prostate enlargement and acceleration of early-stage prostate cancer. The anabolic effects obtained to date from testosterone replacement have been relatively modest, especially in older men. Our hypothesis is that combined treatment with a higher-than-replacement dose of testosterone and a 5- reductase inhibitor will produce substantial anabolic effects, while preventing testosterone-induced prostate enlargement and possibly other adverse effects.

We plan to investigate the efficacy and safety of combined treatment with testosterone and finasteride in older hypogonadal male veterans by conducting a 12-month randomized, placebo-controlled trial. We will administer a higher-than-replacement dose of testosterone plus the 5- reductase inhibitor finasteride to a group of hypogonadal, but otherwise healthy older men. We will determine whether this treatment is a safe and effective means to increase muscle mass and strength. Men aged 60 to 80, with circulating total testosterone 300 ng/dL or bioavailable testosterone 70 ng/dL, will be treated with 125 mg testosterone enanthate/week 5 mg finasteride/day for 1 year. We will assess the effects on body composition, 1- repetition maximum (1-RM) strength, grip strength, functional reach, bone mineral density, mood, cognition, hematopoiesis and prostate volume. We have chosen a moderately high dose of testosterone that may cause some adverse effects. We predict that finasteride will not block the anabolic effects of testosterone, but will block any prostate enlargement or symptoms and possibly other adverse effects as well.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years males
* Primary care at the Malcolm Randall VA Medical Center in Gainesville, Florida.
* Consenting subjects who have a morning (between 6:00 AM and 10:00 AM) serum total testosterone 300 ng/dL or bioavailable testosterone concentration 70 ng/dL and no exclusion criteria will be randomized to receive either testosterone or placebo.

Exclusion Criteria:

* Subjects with cognitive impairment will be identified by the Mini-Cog test and excluded. The Mini-Cog has high sensitivity and specificity for cognitive impairment, and is not affected by level of education.
* We will also exclude subjects with receptive aphasia, or a contraindication to testosterone replacement (i.e., history of or active prostate or breast cancer, severe benign prostatic hyperplasia as assessed by elevated American Urologic Association Symptom Index (AUASI) score > 25), congestive heart failure (Class 3 or 4), sleep apnea syndrome, polycythemia (Hct > 55%), or prostate specific antigen (PSA) > 2.6 ng/mL) will be excluded.
* Obese subjects (BMI > 35) will also be excluded.
* Subjects currently receiving testosterone supplementation or subjects who have an allergy to testosterone will also be excluded.
* Subjects previously receiving testosterone replacement therapy must be off such medication for at least four weeks.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-01; Primary Completion 2012-03 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Borst, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

REFERENCES:
- [Result] Yarrow JF, Beck DT, Conover CF, Beggs LA, Goldberger BA, Borst SE. Invalidation of a commercially available human 5alpha-dihydrotestosterone immunoassay. Steroids. 2013 Dec 11;78(12-13):1220-5. doi: 10.1016/j.steroids.2013.08.013. Epub 2013 Sep 6. PMID 24012740
- [Result] Borst SE, Yarrow JF, Conover CF, Nseyo U, Meuleman JR, Lipinska JA, Braith RW, Beck DT, Martin JS, Morrow M, Roessner S, Beggs LA, McCoy SC, Cannady DF 2nd, Shuster JJ. Musculoskeletal and prostate effects of combined testosterone and finasteride administration in older hypogonadal men: a randomized, controlled trial. Am J Physiol Endocrinol Metab. 2014 Feb 15;306(4):E433-42. doi: 10.1152/ajpendo.00592.2013. Epub 2013 Dec 10. PMID 24326421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between 7/2/2007 and 10/13/2010. Subjects responded to letters mailed to male patients aged 60 years or more who were seen at VA clinics.
Pre-assignment Details: Subjects were excluded if they failed brief cognitive testing (MiniCog), if serum testosterone > 300 ng/dL or less and bio-testosterone > 70 ng/dL, congestive heart failure, sleep apnea, hematocrit (HCT) > 49%, prostate specific antigen (PSA) > 2.6 ng/ml, were taking coumadin or had orthopedic limitations.
Groups:
- Arm 1: testosterone enanthate
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Collection of 3-day food logs with counseling of subjects : subject weighs food portions and completes food log, once/3 months, for 18 months (including 6-month follow-up. Counseling will be healthy ways to increase protein intake, if needed.
- Arm 2: finasteride
  Collection of 3-day food logs with counseling of subjects : subject weighs food portions and completes food log, once/3 months, for 18 months (including 6-month follow-up. Counseling will be healthy ways to increase protein intake, if needed.
  Finasteride : 5 mg, oral, once/day, for 52 weeks
- Arm 3: testosterone enanthate + finasteride
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Finasteride : 5 mg, oral, once/day, for 52 weeks
  Collection of 3-day food logs with counseling of subjects : subject weighs food portions and completes food log, once/3 months, for 18 months (including 6-month follow-up. Counseling will be healthy ways to increase protein intake, if needed.
- Arm 4: placebo
  Collection of 3-day food logs with counseling of subjects : subject weighs food portions and completes food log, once/3 months, for 18 months (including 6-month follow-up. Counseling will be healthy ways to increase protein intake, if needed.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 14 | 13 | 17 | 16
Completed | 7 | 8 | 13 | 12
Not Completed | 7 | 5 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Men aged over 60 with serum testosterone 300 ng/dL or biotestosterone 70 ng/dL or less were recruited
Groups:
- Testosterone Vehicle: 125 mg testosterone enanthate/week i.m. daily placebo pill
- Vehicle Finasteride: weekly vehicle injection 5 mg finasteride/day p.o.
- Testosterone Finasteride: 125 mg testosterone enanthate/week i.m. 5 mg finasteride/day p.o.
- Vehicle Placebo: weekly vehicle injection daily placebo pill
- Total: Total of all reporting groups
Arm/Group | Testosterone Vehicle | Vehicle Finasteride | Testosterone Finasteride | Vehicle Placebo | Total
Number analyzed (Participants) | 14 | 13 | 17 | 16 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (8.0) | 69.5 (9.2) | 64.2 (4.8) | 70.8 (9.7) | 68.25 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 14 | 13 | 17 | 16 | 60

OUTCOME MEASURES:

1. Primary Outcome: 1 Repetition Maximum (1-RM) Strength Testing
Description: 1-RM strength testing for 5 exercises will be performed using dynamic resistance exercise machines. Testing will be performed before treatment (baseline), at 3, 6, 9 and 12 months after treatment.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Population: per protocol
Measure: Mean (Standard Error); unit: kg
Groups:
- Arm 1: testosterone enanthate
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Measurement of leg press strength, 1-RM
- Arm 2: finasteride
  Measurement of leg press strength, 1-RM Finasteride : 5 mg, oral, once/day, for 52 weeks
- Arm 3: testosterone enanthate + finasteride
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Finasteride : 5 mg, oral, once/day, for 52 weeks
  Measurement of leg press strength, 1-RM
- Arm 4: placebo
  Measurement of leg press strength, 1-RM
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 14 | 13 | 17 | 16
kg
  leg press baseline Kg | 129.1 (9.08) | 109.4 (7.87) | 137.2 (5.8) | 118.8 (8.825)
  leg press 3-months change kg | 9.192 (1.978) | -1.34 (3.126) | 9.679 (3.16) | -2.44 (2.22)
  leg press 6-months change kg | 10.227 (1.66) | -1.136 (4.095) | 13.778 (4.1) | 2.727 (3.66)
  leg press 9-months change kg | 14.416 (2.63) | -5.55 (4.95) | 10.49 (3.1) | 2.02 (2.636)
  leg press 12-months change kg | 14.773 (7.03) | 0 (2.629) | 12.5 (3.88) | 1.515 (3.47)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; The studies was powered for 1-RM strength based on a 1.18-alpha increase reported in the literature; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The difference in means and p value are for 12 months (using data from all time points to make the calculation). We tested the effect of testosterone ([T-placebo plus T-finasteride] vs. [vehicle-placebo plus vehicle-finasteride]); Mean Difference (Net) = 12.9, 95% CI 2-sided [7.86 to 18.0], Standard Deviation 2.57 — mean difference is for subjects reveiving testosterone (groups T and T/F) vs. subjects not receiving testosterone (F and Placebo)

2. Secondary Outcome: Grip Strength kg
Description: Grip strength in the dominant arm will be measured by using a dynamometer. Testing will be performed at baseline, after 3, 6, 9 and 12 months of treatment.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Measure: Mean (Standard Error); unit: kg
Groups:
- Testosterone Vehicle: testosterone enanthate
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  grip strength measure on a dynamometer
- Vehicle Finasteride; Testosterone Finasteride; Vehicle Placebo: grip strength measure on a dynamometer
Arm/Group | Testosterone Vehicle | Vehicle Finasteride | Testosterone Finasteride | Vehicle Placebo
Number analyzed (Participants) | 14 | 13 | 17 | 16
kg
  grip strength baseline kg | 17.0 (1.23) | 16.9 (1.28) | 18.2 (0.513) | 17.472 (0.8522)
  change grip strength 3 month kg | 1.66 (.427) | -0.045 (0.485) | 0.485 (0.447) | 0.212 (0.44)
  change grip strength 6 month kg | 2.02 (0.482) | 0.812 (1.357) | 1.00 (0.589) | -0.035 (0.411)
  change grip strength 9 month kg | 1.558 (0.505) | 1.25 (0.555) | 1.331 (0.399) | 0.152 (0.415)
  change grip strength 12 month kg | 1.909 (0.249) | 1.477 (0.211) | 1.174 (0.302) | 0.72 (0.342)
Statistical Analysis 1: Comparison: Testosterone Vehicle vs Vehicle Finasteride vs Testosterone Finasteride vs Vehicle Placebo; The study was not powered on grip strength. We employed 2x2 analysis to determine effects of testosterone, finasteride and interaction; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.77, 95% CI 2-sided [0.16 to 1.31], Standard Deviation 0.311

3. Secondary Outcome: Lumbar Spine L2-L4 Bone Mineral Density
Description: Dual x-ray absorptiometry (DXA): We will assess bone mineral density (BMD) and body composition using a fan-bean densitometer (Lunar Prodigy, General Electric Medical Systems).
Time Frame: baseline, 12 months
Measure: Mean (Standard Error); unit: gm/cc
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 14 | 13 | 17 | 16
gm/cc
  L2-L4 spine BMD baseline gm/cc | 1.03 (0.041) | 1.02 (0.032) | 0.99 (0.0167) | 1.07 (0.045)
  change L2-L4 spine BMD 12 month gm/cc | 0.049 (0.017) | 0.002 (0.006) | 0.053 (0.017) | -0.020 (0.011)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; The study was not powered on lumbar spine bone mineral density. We employed a 2x2 analysis for effects ot testosterone, finasteride and interaction; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 4.19, 95% CI 2-sided [1.95 to 6.43], Standard Deviation 1.142

4. Secondary Outcome: Geriatric Depression Scale
Description: Geriatric Depression Scale (GDS): This 15-item, yes/no questionnaire will be administered at baseline, after 3, 6, 9 and 12 months of treatment.
  The minimum score is 0 = no depressive symptoms The maximum score is 15 = a very high level of depressive symptoms
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Testosterone Vehicle; Vehicle Finasteride; Testosterone Finasteride; Vehicle Placebo: Geriatric Depression Scale (GDS): This 15-item, yes/no questionnaire will be administered at baseline, after 3, 6, 9 and 12 months of treatment and at follow-up.
Arm/Group | Testosterone Vehicle | Vehicle Finasteride | Testosterone Finasteride | Vehicle Placebo
Number analyzed (Participants) | 14 | 13 | 17 | 16
units on a scale
  depression baseline | 2.38 (0.49) | 3.08 (1.09) | 4.93 (2.76) | 2.13 (0.48)
  depression 3 months | 1.80 (0.49) | 2.90 (1.24) | 3.23 (0.86) | 1.67 (0.3)
  depression 6 months | 1.5 (0.48) | 2.22 (1.30) | 5.0 (1.33) | 1.62 (0.5)
  depression 9 months | 0.88 (0.23) | 1.89 (0.99) | 3.69 (1.07) | 2.92 (0.94)
  depression 12 months | 3.33 (1.38) | 2.88 (1.42) | 3.73 (1.18) | 1.83 (0.373)
Statistical Analysis 1: Comparison: Testosterone Vehicle vs Vehicle Finasteride vs Testosterone Finasteride vs Vehicle Placebo; The study is was not powered for score on Geriatric Depression Scale; Test type: Superiority or Other; p = 0.037, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.737, 95% CI 2-sided [-1.41 to -0.064], Standard Error of Mean 0.343

5. Secondary Outcome: 30 Minute Recall Portion of Rey Osterrieth Complex Figure (ROCF) Test
Description: Rey Osterrieth Complex Figure (ROCF) test is a widely used standardized neuropsychological test for assessing visuospatial constructional functions, visuographic memory, and some aspects of planning.
  The drawing is scored by a blinded neuropsychologist on a scale of 0 to 30 with 30 representing a perfect drawing.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Arm 1: testosterone enanthate
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  30 minute recall portion of Rey Osterrieth Complex Figure (ROCF) test
- Arm 2: finasteride
  30 minute recall portion of Rey Osterrieth Complex Figure (ROCF) test Finasteride : 5 mg, oral, once/day, for 52 weeks
- Arm 3: testosterone enanthate + finasteride
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Finasteride : 5 mg, oral, once/day, for 52 weeks
  30 minute recall portion of Rey Osterrieth Complex Figure (ROCF) test
- Arm 4: placebo
  30 minute recall portion of Rey Osterrieth Complex Figure (ROCF) test
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 14 | 13 | 17 | 16
units on a scale
  Rey baseline | 12.42 (1.46) | 13.54 (1.36) | 12.82 (0.92) | 12.8 (1.58)
  Rey 3 month | 16.68 (2.25) | 12.85 (1.57) | 16.27 (1.6) | 12.5 (1.5)
  Rey 6 month | 15.76 (2.6) | 16.17 (2.04) | 17.38 (1.55) | 14 (2.7)
  Rey 9 month | 15.25 (3.06) | 15.17 (2.27) | 18.08 (1.39) | 15.55 (2.45)
  Rey 12 month | 16.86 (2.91) | 15 (2.56) | 19.27 (1.98) | 16.45 (2.77)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; The study was not powered for 30-minute recall on Rey figure test; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.871, 95% CI 2-sided [0.699 to 5.04], Standard Error of Mean 1.108

6. Secondary Outcome: Trail-Making Test, Part A
Description: Trail-Making Test, Part A: is a standardized test of cognitive function which specifically assesses working memory, visual processing, visual spatial skills, selective and divided attention, and psychomotor coordination. the test is scored as seconds required to successful completion of the task with a lower score representing better performance. The mean score on test is 30.75 second with a standard deviation of 16.27.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Measure: Mean (Standard Error); unit: sec
Groups:
- Arm 1: testosterone enanthate
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Trail Making Test A
- Arm 2: finasteride
  Trail Making Test A Finasteride : 5 mg, oral, once/day, for 52 weeks
- Arm 3: testosterone enanthate + finasteride
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Finasteride : 5 mg, oral, once/day, for 52 weeks
  Trail Making Test A
- Arm 4: placebo
  Trail Making Test A
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 14 | 13 | 17 | 16
sec
  Trails A baseline | 37.59 (3.58) | 46.42 (3.61) | 36.65 (2.24) | 44.0 (6.76)
  Trails A 3 months | 38.5 (5.24) | 42.1 (5.59) | 33.53 (1.83) | 44.33 (7.12)
  Trails A 6 months | 32.9 (3.91) | 39.0 (5.55) | 31.2 (2.1) | 36.92 (5.21)
  Trails A 9 months | 31.0 (4.48) | 38.56 (4.37) | 29.07 (1.73) | 43.17 (12.97)
  Trails A 12 months | 29.17 (6.47) | 40.0 (5.48) | 32.5 (2.98) | 43.75 (13.26)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; The study was not powered for score on Trials A test; Test type: Superiority or Other; p = 0.779, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.642, 95% CI 2-sided [-5.095 to 3.811], Standard Error of Mean 2.272

7. Secondary Outcome: Benton Judgment of Line Orientation Test
Description: Benton Judgment of Line Orientation Test is a standardized test with 30 items that is specific for visual spatial cognition. Tests will be administered at baseline, after 3, 6, 9 and 12 months of treatment.
  The minimum score is 0, indicating low visual spatial cognition. The maximum score is 30, indicating high visual spatial cognition
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Arm 1: testosterone enanthate
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Benton Test -Judgment of Line Orientation
- Arm 2: finasteride
  Benton Test -Judgment of Line Orientation
  Finasteride : 5 mg, oral, once/day, for 52 weeks
- Arm 3: testosterone enanthate + finasteride
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Finasteride : 5 mg, oral, once/day, for 52 weeks
  Benton Test -Judgment of Line Orientation
- Arm 4: placebo
  Benton Test -Judgment of Line Orientation
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 14 | 13 | 17 | 16
units on a scale
  Benton baseline | 24.54 (1.26) | 24.39 (0.80) | 25.88 (0.92) | 24.69 (1.23)
  Benton 3 months | 25.00 (0.73) | 25.40 (1.38) | 25.07 (1.09) | 25.67 (1.17)
  Benton 6 months | 25.90 (1.18) | 25.11 (1.33) | 26.0 (0.79) | 25.08 (1.26)
  Benton 9 months | 25.38 (1.48) | 23.89 (1.23) | 25.79 (0.81) | 24.92 (1.75)
  Benton 12 months | 25.67 (0.80) | 25.5 (1.12) | 26.17 (0.77) | 24.08 (1.88)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; The study was not powered for score on Benton test; Test type: Superiority or Other; p = 0.433, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.587, 95% CI 2-sided [-0.869 to 2.043], Standard Error of Mean 0.743

8. Secondary Outcome: Hematocrit
Description: Hematocrit was assessed as a part of routine blood analysis at the indicated time points.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Measure: Mean (Standard Error); unit: % volume
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 14 | 13 | 17 | 16
% volume
  hematocrit baseline % | 42.6 (0.833) | 41.2 (1.042) | 42.0 (0.7) | 40.3 (0.975)
  change hematocrit 3 months % | 3.6 (1.007) | 0.611 (1.143) | 4.593 (0.627) | -0.06 (0.44)
  change hematocrit 6 months % | 4.044 (0.94) | 0.557 (0.758) | 4.331 (0.7264) | 0.514 (0.396)
  change hematocrit 9 months % | 4.071 (1.303) | 0.63 (1.36) | 3.38 (0.6622) | -0.155 (0.52)
  change hematocrit 12 months % | 5.22 (0.8498) | -1.175 (0.984) | 4.173 (0.8498) | -0.192 (0.667)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; This study was powered for hematocrit based on literature report that testosterone > 2 alpha increase in hematocrit; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 4.13, 95% CI 2-sided [3.07 to 5.18], Standard Deviation 0.540

9. Secondary Outcome: Dietary Protein Intake
Description: Dietary protein intake will be assessed using a 3-day food log and subjects will be counseled to increase protein intake if needed using the guide "Healthy Ways to Eat More Protein".
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Measure: Mean (Standard Error); unit: gm/body weight (kg)
Groups:
- Arm 1: testosterone enanthate
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Daily dietary protein intake (gm/kg body weight) derived from 3-day food log
- Arm 2: finasteride
  Finasteride : 5 mg, oral, once/day, for 52 weeks
  Daily dietary protein intake (gm/kg body weight) derived from 3-day food log
- Arm 3: testosterone enanthate + finasteride
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Finasteride : 5 mg, oral, once/day, for 52 weeks
  Daily dietary protein intake (gm/kg body weight) derived from 3-day food log
- Arm 4: placebo
  Daily dietary protein intake (gm/kg body weight) derived from 3-day food log
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 14 | 13 | 17 | 16
gm/body weight (kg)
  protein intake baseline | 0.97 (0.10) | 1.06 (0.08) | 0.99 (0.13) | 1.00 (0.06)
  protein intake 3 months | 0.87 (0.16) | 0.94 (0.15) | 1.49 (0.18) | 1.12 (0.16)
  protein intake 6 months | 0.74 (0.07) | 1.27 (0.49) | 1.05 (0.18) | 0.93 (0.18)
  protein intake 9 months | 1.15 (0.08) | 1.20 (0.30) | 1.26 (0.30) | 0.82 (0.09)
  protein intake 12 months n = 1,1,2,5 | 1.18 (NA) — insufficient data for standard deviation | 0.74 (NA) — insufficient data for standard deviation | 1.39 (0.60) | 1.05 (0.18)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; The study was not powered for dietary protein intake; Test type: Superiority or Other; p = 0.6219, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.1419, 95% CI 2-sided [-0.353 to 6.37], Standard Error of Mean 0.2529

10. Secondary Outcome: Transrectal Ultrasound Sizing of Prostate
Description: Transrectal ultrasound sizing of prostate will be performed using the B&K Diagnostic System 3535, with 7 mega hertz transrectal probe at baseline and after 6 and 12 months of treatment.
Time Frame: baseline, 6 month, 12 months
Measure: Mean (Standard Error); unit: cc
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 14 | 13 | 17 | 16
cc
  postate volume baseline cc | 26.4 (2.33) | 29.7 (3.395) | 37.1 (4.379) | 36.9 (3.9)
  change prostate volume 6 months cc | 7.626 (1.703) | -1.984 (4.31) | -3.927 (2.25) | -1.474 (3.147)
  change prostate volume 12 months cc | 11.42 (3.9) | -4.93 (3.3) | -1.72 (1.596) | -2.891 (2.57)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; The study was powered for prostate volume based on a literature report that testosterone increases prostate volume 1.85 alpha per year. We employed a 2x2 analysis for effects of testosterone, finasteride and interaction; Test type: Superiority or Other; p = 0.0051, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 5.33, 95% CI 2-sided [1.73 to 8.94], Standard Deviation 1.83

11. Secondary Outcome: Life Satisfaction
Description: Life Satisfaction: is a written test of psychological well-being that will be performed at baseline, after 3, 6, 9 and 12 months of treatment. This is a 20-point scale, with a possible range of scores from 0 to 20. A higher score represents greater life satisfaction.
Time Frame: baseline, 3 months, 6 months, 9 months, 12 months
Measure: Mean (Standard Error); unit: points
Groups:
- Arm 1: testosterone enanthate
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Life Satisfaction A
- Arm 2: finasteride
  Finasteride : 5 mg, oral, once/day, for 52 weeks
  Life Satisfaction A
- Arm 3: testosterone enanthate + finasteride
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Finasteride : 5 mg, oral, once/day, for 52 weeks
  Life Satisfaction A
- Arm 4: placebo
  Life Satisfaction A
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 14 | 13 | 17 | 16
points
  Life Satisfaction A baseline | 13.83 (1.01) | 12.08 (1.65) | 11.35 (1.11) | 12.69 (1.08)
  Life Satisfaction A 3 months | 12.67 (0.76) | 12.11 (2.00) | 12.27 (1.33) | 14.13 (0.91)
  Life Satisfaction A 6 months | 13.70 (1.05) | 14.44 (1.65) | 11.20 (1.59) | 13.54 (1.26)
  Life Satisfaction A 9 months | 14.75 (1.03) | 13.44 (1.39) | 11.57 (1.35) | 13.17 (1.48)
  Life Satisfaction A 12 months | 15.17 (1.11) | 12.5 (1.91) | 12.17 (1.80) | 13.83 (1.38)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; The study was not powered for score on Lif Satisfaction A test; Test type: Superiority or Other; p = 0.196, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -.868, 95% CI 2-sided [-3.434 to 1.698], Standard Error of Mean 0.668

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Arm 1: testosterone enanthate
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
- Arm 2: finasteride
  Finasteride : 5 mg, oral, once/day, for 52 weeks
- Arm 3: testosterone enanthate + finasteride
  Testosterone Enanthate : 125 mg, i.m. injection, once/week, for 52 weeks
  Finasteride : 5 mg, oral, once/day, for 52 weeks
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Serious Adverse Events (participants affected / at risk) | 3/14 | 2/13 | 0/17 | 1/16
Other Adverse Events (participants affected / at risk) | 2/14 | 1/13 | 2/17 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=14) | Arm 2 (N=13) | Arm 3 (N=17) | Arm 4 (N=16)
Paget's disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
stroke (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
sleep apnea (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — 83-year old subject did not show up for visits. We learned from the newspaper that he had dies, but did not learn the cause of death.
surgery for pre-existing heart condition (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subject had a pre-existing heart condition that did not preclude participation and thought that he might have surgery after the study. it was then decided to schedule the surgery sooner, so participation in the study stopped.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=14) | Arm 2 (N=13) | Arm 3 (N=17) | Arm 4 (N=16)
elevated prostate specific antigen (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — elevate PSA was defined as 2.6 or greater for study purposes
urinary symptoms (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — urinary symptoms defined as an increased score on urinary symptom questionaire
elevated hematocrit (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — elevated hematocrit was defined as 54 or greater

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less